CLINICAL TRIAL: NCT01591720
Title: Effectiveness Testing of a Tailored Internet-delivered Cognitive Behaviour Therapy Treatment for Symptoms of Depression, Anxiety and Comorbid Problems
Brief Title: Tailored Internet-delivered Cognitive Behaviour Therapy in Primary Care
Acronym: TAYLOR2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Gerhard Andersson, Professor of Clinical Psychology, Linkoeping University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GA-VR-DEP-2
Record Dates: First submitted 2012-04-18; First posted 2012-05-04 (Estimated); Last update posted 2012-05-04 (Estimated); Status verified 2012-05

CONDITIONS: Depression; Anxiety Disorders
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tailored Internet-delivered CBT (Experimental): The intervention is delivered within a primary care clinic.
  Interventions: Behavioral: Tailored Internet-based CBT for depression and anxiety

INTERVENTIONS:
Behavioral: Tailored Internet-based CBT for depression and anxiety — This Internet-based CBT intervention contains 8-10 text-based self-help modules in which 4 modules are fixed (the first three and the last) and the rest are "prescribed" following the diagnostic interview. These modules contain material on panic disorder, social phobia, stress management, assertiveness training, concentration, relaxation among other things.

SUMMARY:
A tailored Internet-based cognitive-behavioural intervention is tested within a primary care clinic. Weekly measures of symptoms of depression and anxiety are obtained. Significant within-group effects are expected.

DETAILED DESCRIPTION:
This Internet-based cognitive-behavioural therapy intervention contains 8-10 text-based self-help modules in which 4 modules are fixed (the first three and the last) and the rest are "prescribed" following the diagnostic interview. These modules contain material on panic disorder, social phobia, stress management, assertiveness training, concentration, relaxation among other things.

The intervention is tested within a primary care clinic. Weekly measures of symptoms of depression and anxiety are obtained.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of depression and anxiety

Exclusion Criteria:

* Severe depression (based on interview)
* Severe psychiatric condition (e.g. psychosis or bipolar disorder)
* Suicidal (measured in diagnostic interview)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2010-09; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire 9 (PHQ-9) | 2 weeks before treatment starts
Patient Health Questionnaire 9 (PHQ-9) | Weekly measures during treatment (for up to 16 weeks)
Patient Health Questionnaire 9 (PHQ-9) | At treatment termination (after a maximum of 16 weeks)
Generalised Anxiety Disorder Assessment 7 (GAD-7) | 2 weeks before treatment starts
Generalised Anxiety Disorder Assessment 7 (GAD-7) | Weekly measures during treatment (for up to 16 weeks)
Generalised Anxiety Disorder Assessment 7 (GAD-7) | At treatment termination (after a maximum of 16 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Andersson, PhD, Principal Investigator — Department of Behavioral Sciences and Learning, Linköping University
Locations (1):
- Linköping University, Department of Behavioral Sciences and Learning, Linköping, Sweden